CLINICAL TRIAL: NCT04350918
Title: Effects Muscle Energy Technique and Static Stretching on Pain Intensity and Functional Disability in Patients With Mechanical Neck Pain: A Randomized Control Study
Brief Title: Muscle Energy Technique and Static Stretching on Pain Intensity and Functional Disability in Patients With Mechanical Neck Pain
Acronym: MET&SSinNckp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Adesola Ojo Ojoawo, Dr and Head of Department, Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OJO/2020/01
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Neck Pain
Keywords: Static stretching, ,; neck pain,; muscle energy techniques; visual analogue scale,; neck disability index
MeSH Terms: conditions — Neck Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Subjects for this study were patients diagnosed of mechanical neck pain in Physiotherapy Outpatient Department of Obafemi Awolowo University Teaching Hospital Complex (OAUTHC), Ile-Ife. Individuals who meet the inclusion criteria were randomly allocated to Muscle Energy Techniques Group and Static Stretching Group using the simple random assignment method without replacement (Fish Bowl).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique (MET) (Experimental): MET Group received 12 treatment sessions of MET (Nagrale et al, 2010) two times a week in addition to conventional physiotherapy. The procedures employ voluntary muscle contractions by the patient in a precisely controlled direction and intensity against a counterforce applied by the Physiotherapist. The technique requires the therapist to provide stabilization to the segment on which the distal aspect of the muscle attaches. A command for anisometric contraction of the muscle is given that causes accessory movement of the joint. Several specific muscle energy techniques are described for the subcranial region of the cervical spine.
  Interventions: Device: Muscle Enery Techniques
- Static stretching (SS) (Experimental): Subjects in SS Group received 12 treatment sessions of static stretching (Dutton et al, 2008) two times a week in addition to conventional physiotherapy.
  Stretching involves the application of manual or mechanical force to elongate structures that have adaptively shortened and are hypo-mobile (Sullivan, 2007) Static stretching involves stretching a muscle to a point of discomfort and holding the stretch for a length of time, followed by a return to normal resting muscle length (Andrews et al, 2004). Muscles of the neck were stretched in especially in side flexion, extension, flexion and side rotation for 10 seconds and was repeated 10 times for a session.
  Interventions: Device: Static Stretching

INTERVENTIONS:
Device: Muscle Enery Techniques — Group of patients that underwent muscle energy technique as a mean of treatment for the complaint
  Other Names: MET
  Arms: Muscle Energy Technique (MET)
Device: Static Stretching — Set of patients that had static stretching technique for the treatment for the complaint
  Other Names: SS
  Arms: Static stretching (SS)

SUMMARY:
Neck pain is becoming increasingly common throughout the world with a considerable impact on individuals, communities, health-care systems and businesses (Hoy et al, 2011).Neck pain is a common problem within our society affecting individual's physical and social functioning considerably and interfering with the patient's daily activities. There is lack of evidence to allow conclusions to be drawn about the effectiveness of MET when compared with stretching exercises for relieving mechanical neck pain. Therefore, this study is designed to examine the effect of MET, static stretching and to compare their effects on pain intensity and functional disability in patient with mechanical neck pain.

DETAILED DESCRIPTION:
This experimental study purposively recruited 24 subjects (male: n=10, female: n = 14) with mechanical neck pain from the Outpatient Physiotherapy Department of the Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife. Subjects were randomly allocated into the MET and SS groups. Subjects in MET group received 6 treatment sessions of Muscle Energy Technique in addition to conventional physiotherapy treatments. Patients in SS group received 6 treatment sessions of Static Stretching in addition to conventional physiotherapy treatments. All subjects were treated twice a week for six weeks. Visual Analogue Scale (VAS) and Neck Disability Index (NDI) were used to assess the pain intensity and functional disability at baseline, 3rd week and 6th week of treatment sessions respectively. Descriptive and Inferential statistics were used to analyse the data. Alpha level was set at < 0.05.

ELIGIBILITY:
Inclusion Criteria:i. Male and female patients with history of mechanical neck pain of more than 3 months

Exclusion Criteria:

* Patients with acute neck pain
* Subjects were excluded if they have neck pain associated with an underlying pathology such as fracture of the cervical spine, neck pain radiating into the arms or upper extremity or associated with headaches or facial pain, malignancy, infections, inflammatory disorders, osteoporosis or cases of disc prolapse.
* Patients with history of surgery of the cervical spine during the previous 12months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | From March 2019 to November 2019, The treatment for each patient was for 6 weeks
  VAS is a one-dimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases (Mc Cormack et al, 1988). pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm) (Aun et al, 1986)

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | From March 2019 to November 2019, The treatment for each patient was for 6 weeks
  The NDI can be scored as a raw score or doubled and expressed as a percent (Vernon, 1991). Each session is scored on a 0 to 5 rating scale, in which zero means 'No Pain' and 5 means 'Worst Imaginable Pain'. All the points can be summarized as a total score. The test can be interpreted as a raw score with a maximum score of 50 or as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Adesola O Ojoawo PhD, Principal Investigator — Head, Department of Medical Rehabilitation, Obafemi Awolowo University Ile Ife; Kayode Ijaduola, Study Chair — Provost, College of Health Sciences, Obafemi Awolowo University
Locations (1):
- Obafemi Awolowo University, Ile-Ife, Osun State, Nigeria